CLINICAL TRIAL: NCT01922089
Title: A Multicenter, Randomized, Double-blind, Parallel Group Study to Assess the Safety and Tolerability of Initiating LCZ696 in Heart Failure Patients Comparing Two Titration Regimens
Brief Title: Safety and Tolerability of Initiating LCZ696 in Heart Failure Patients
Acronym: TITRATION
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLCZ696B2228; 2013-001835-33 (EudraCT Number)
Record Dates: First submitted 2013-08-12; First posted 2013-08-14 (Estimated); Results first posted 2015-10-15 (Estimated); Last update posted 2015-10-15 (Estimated); Status verified 2015-09

CONDITIONS: Heart Failure With Reduced Ejection Fraction
Keywords: Heart failure, reduced ejection fraction, LCZ696, titration, safety, tolerability
MeSH Terms: conditions — Heart Failure | interventions — sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- LCZ696 Condensed (Experimental): Up-titration to LCZ696 200 mg twice daily (bid) over 3 weeks
  Interventions: Drug: LCZ696
- LCZ696 Conservative (Experimental): Up-titration to LCZ696 200 mg bid over 6 weeks
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 50 mg/100 mg/200 mg bid

SUMMARY:
The purpose of this study is to assess the safety and tolerability of initiating LCZ696 in heart failure patients with reduced ejection fraction (HF-rEF) using conservative (reaching target dose over 6 weeks) and condensed (reaching target dose over 3 weeks) up-titration regimens.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years; CHF with New York Heart Association class II-IV; left ventricular ejection fraction ≤ 35%; on beta blockers

Exclusion Criteria:

* Potassium > 5.2 mmol/l; estimated glomerular filtration rate < 30 ml/min/1.73 m2; systolic blood pressure <100 mmHg or > 180 mmHg; history of intolerance to recommended target doses of angiotensin converting enzyme inhibitors or angiotensin receptor blockers

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 498 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (92):
- United States (21):
  - Novartis Investigative Site, Anchorage, Alaska
  - Novartis Investigative Site, Gilbert, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Anaheim, California
  - Novartis Investigative Site, Torrance, California
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Chiefland, Florida
  - Novartis Investigative Site, Aurora, Illinois
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Evansville, Indiana
  - Novartis Investigative Site, Slidell, Louisiana
  - Novartis Investigative Site, Minneapolis, Minnesota
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Buffalo, New York
  - Novartis Investigative Site, Laurelton, New York
  - Novartis Investigative Site, Marion, Ohio
  - Novartis Investigative Site, Oak Ridge, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Livingston, Texas
  - Novartis Investigative Site, Tacoma, Washington
- Bulgaria (4):
  - Novartis Investigative Site, Gabrovo, Bulgaria
  - Novartis Investigative Site, Plovdiv, Bulgaria
  - Novartis Investigative Site, Smolyan, Bulgaria
  - Novartis Investigative Site, Sofia
- Finland (2):
  - Novartis Investigative Site, Jyväskylä
  - Novartis Investigative Site, Tampere
- Germany (18):
  - Novartis Investigative Site, Bad Krozingen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Buch
  - Novartis Investigative Site, Dietzenbach
  - Novartis Investigative Site, Ebersbach
  - Novartis Investigative Site, Frankfurt
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Haßloch
  - Novartis Investigative Site, Huy / OT Anderbeck
  - Novartis Investigative Site, Ingelheim
  - Novartis Investigative Site, Kelkheim
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Leipzig
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mühlheim
  - Novartis Investigative Site, Siegen
  - Novartis Investigative Site, Straubing
  - Novartis Investigative Site, Würzburg
- Hungary (6):
  - Novartis Investigative Site, Budapest
  - Novartis Investigative Site, Debrecen
  - Novartis Investigative Site, Mosonmagyaróvár
  - Novartis Investigative Site, Nyiregyháza
  - Novartis Investigative Site, Pécs
  - Novartis Investigative Site, Székesfehérvár
- Italy (10):
  - Novartis Investigative Site, Aosta, AO
  - Novartis Investigative Site, Cortona, AR
  - Novartis Investigative Site, Bergamo, BG
  - Novartis Investigative Site, Bologna, BO
  - Novartis Investigative Site, Cona, FE
  - Novartis Investigative Site, Albano Laziale, RM
  - Novartis Investigative Site, Roma, RM
  - Novartis Investigative Site, Sassari, SS
  - Novartis Investigative Site, Vittorio Veneto, TV
  - Novartis Investigative Site, San Daniele del Friuli, UD
- Novartis Investigative Site, San Juan, Puerto Rico
- Slovakia (8):
  - Novartis Investigative Site, Brezno, Slovak Republic
  - Novartis Investigative Site, Nitra, Slovak Republic
  - Novartis Investigative Site, Svidník, Slovak Republic
  - Novartis Investigative Site, Bratislava, Slovakia
  - Novartis Investigative Site, Košice, Slovakia
  - Novartis Investigative Site, Lučenec, Slovakia
  - Novartis Investigative Site, Nové Zámky, Slovakia
  - Novartis Investigative Site, Trebišov, Slovakia
- Spain (8):
  - Novartis Investigative Site, Almería, Andalusia
  - Novartis Investigative Site, Málaga, Andalusia
  - Novartis Investigative Site, Sanlúcar de Barrameda, Andalusia
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Villamartín, Cadiz
  - Novartis Investigative Site, Barcelona, Catalonia
  - Novartis Investigative Site, A Coruña, Galicia
  - Novartis Investigative Site, Madrid, Madrid
- Turkey (Türkiye) (5):
  - Novartis Investigative Site, Istanbul, Turkey
  - Novartis Investigative Site, Haydarpasa/Istanbul
  - Novartis Investigative Site, Kocaeli
  - Novartis Investigative Site, Mersin
  - Novartis Investigative Site, Sivas
- United Kingdom (9):
  - Novartis Investigative Site, Dorchester, Dorset
  - Novartis Investigative Site, Saint Leonards-on-Sea, East Sussex
  - Novartis Investigative Site, Oldham, Lancashire
  - Novartis Investigative Site, Gateshead, Tyne and Wear
  - Novartis Investigative Site, Bath
  - Novartis Investigative Site, Bradford
  - Novartis Investigative Site, Coventry
  - Novartis Investigative Site, Harrow
  - Novartis Investigative Site, Nuneaton

REFERENCES:
- [Derived] Senni M, McMurray JJV, Wachter R, McIntyre HF, Anand IS, Duino V, Sarkar A, Shi V, Charney A. Impact of systolic blood pressure on the safety and tolerability of initiating and up-titrating sacubitril/valsartan in patients with heart failure and reduced ejection fraction: insights from the TITRATION study. Eur J Heart Fail. 2018 Mar;20(3):491-500. doi: 10.1002/ejhf.1054. Epub 2017 Nov 22. PMID 29164797
- [Derived] Senni M, McMurray JJ, Wachter R, McIntyre HF, Reyes A, Majercak I, Andreka P, Shehova-Yankova N, Anand I, Yilmaz MB, Gogia H, Martinez-Selles M, Fischer S, Zilahi Z, Cosmi F, Gelev V, Galve E, Gomez-Doblas JJ, Nociar J, Radomska M, Sokolova B, Volterrani M, Sarkar A, Reimund B, Chen F, Charney A. Initiating sacubitril/valsartan (LCZ696) in heart failure: results of TITRATION, a double-blind, randomized comparison of two uptitration regimens. Eur J Heart Fail. 2016 Sep;18(9):1193-202. doi: 10.1002/ejhf.548. Epub 2016 May 12. PMID 27170530

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LCZ696 Condensed | LCZ696 Conservative
Started | 247 | 251
Safety Set | 246 | 251
Completed | 208 | 221
Not Completed | 39 | 30
Not completed — Adverse Event | 18 | 13
Not completed — Protocol Deviation | 10 | 7
Not completed — Withdrawal by Subject | 3 | 4
Not completed — administrative problems | 4 | 1
Not completed — Physician Decision | 2 | 3
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LCZ696 Condensed | LCZ696 Conservative | Total
Number analyzed (Participants) | 247 | 251 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (11.86) | 63.8 (10.94) | 64.0 (11.39)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 50 | 106
  Male | 191 | 201 | 392

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Hypotension, Renal Dysfunction, Hyperkalemia and Angioedema and by Renin-Angiotensin-Aldosterone System (RAAS) Stratum (High vs. Low)
Description: Participants experiencing hypotension, renal dysfunction, hyperkalemia and angioedema and by Renin-Angiotensin-Aldosterone System (RAAS) stratum (high vs. low) High RAAS stratum Patients receiving > 160 mg of valsartan or > 10 mg total daily dose of enalapril, or equivalent doses of other ARBs/ACEIs, respectively, at screening Low RAAS stratum: Patients receiving ≤ 160 mg of valsartan or ≤ 10 mg total daily dose of enalapril, or equivalent doses of other ARBs/ACEIs, respectively, at screening. This stratum also included patients who were not on an ACEI or an ARB 4 weeks prior to screening (i.e., ACEI/ARB-naïve patients)
Time Frame: 12 weeks
Population: Full Analysis Set (FAS) consisted of all randomized patients with the exception of mis-randomized patients who had not received the study drug, but had been inadvertently randomized into the study. Following the intent-to-treat principle, patients were analyzed according to the treatment to which they were assigned at randomization.
Measure: Number; unit: participants
Arm/Group | LCZ696 Condensed | LCZ696 Conservative
Number analyzed (Participants) | 247 | 251
participants
  Hypotension High RAAS (n=120, 127) | 5 | 7
  Hypotension Low RAAS (n=127, 124) | 19 | 14
  Hypotension ALL | 24 | 21
  Renal Dysfunction High RAAS (n=120, 127) | 5 | 9
  Renal Dysfunction Low RAAS (n=127, 124) | 13 | 10
  Renal Dysfunction ALL | 18 | 19
  Hyperkalemia High RAAS (n=120, 127) | 8 | 5
  Hyperkalemia Low RAAS (n=127, 124) | 11 | 6
  Hyperkalemia ALL | 19 | 11
  Angioedema High RAAS (n=120, 127) | 0 | 1
  Angioedema Low RAAS (n=127, 124) | 0 | 1
  Angioedema ALL | 0 | 2

2. Secondary Outcome: Number of Participants Who Achieved Treatment Success Over the 12 Weeks and by Renin-Angiotensin-Aldosterone System (RAAS) Stratum (High vs. Low)
Description: Treatment success was defined as the number of participants who achieved and maintained LCZ696 200 mg bid without any dose interruption or down-titration over 12 weeks and by Renin-Angiotensin-Aldosterone System (RAAS) stratum (high vs. low) High RAAS stratum Patients receiving > 160 mg of valsartan or > 10 mg total daily dose of enalapril, or equivalent doses of other ARBs/ACEIs, respectively, at screening Low RAAS stratum: Patients receiving ≤ 160 mg of valsartan or ≤ 10 mg total daily dose of enalapril, or equivalent doses of other ARBs/ACEIs, respectively, at screening. This stratum also included patients who were not on an ACEI or an ARB 4 weeks prior to screening (i.e., ACEI/ARB-naïve patients)
Time Frame: 12 weeks
Population: Evaluable patients in FAS with the exception of misrandomized patients who didn't received drug, but had been randomized into the study, excluding patients who discontinued the study prior to completion of 12 wks. Following the intent-to-treat principle, patients were analyzed according to the treatment to which they were assigned at randomization.
Measure: Number; unit: participants
Arm/Group | LCZ696 Condensed | LCZ696 Conservative
Number analyzed (Participants) | 230 | 236
participants
  High RAAS (n=109,117) | 90 | 98
  Low RAAS (n=121,119) | 89 | 101
  ALL (n=230,236) | 179 | 199

3. Secondary Outcome: Number of Participants Who Tolerated Study Medication for at Least the Last Two Weeks of the Study and by Renin-Angiotensin-Aldosterone System (RAAS) Stratum (High vs. Low).
Description: Tolerability was assessed as the number of participants who achieved LCZ696 200 mg bid and maintained this dose for at least 2 weeks before study completion, regardless of previous dose interruption or down-titration and by Renin-Angiotensin-Aldosterone System (RAAS) stratum (high vs. low) High RAAS stratum Patients receiving > 160 mg of valsartan or > 10 mg total daily dose of enalapril, or equivalent doses of other ARBs/ACEIs, respectively, at screening Low RAAS stratum: Patients receiving ≤ 160 mg of valsartan or ≤ 10 mg total daily dose of enalapril, or equivalent doses of other ARBs/ACEIs, respectively, at screening. This stratum also included patients who were not on an ACEI or an ARB 4 weeks prior to screening (i.e., ACEI/ARB-naïve patients)
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | LCZ696 Condensed | LCZ696 Conservative
Number analyzed (Participants) | 230 | 236
participants
  High RAAS (n=109,117) | 94 | 103
  Low RAAS (n=121,119) | 97 | 103
  ALL (n=230,236) | 191 | 206

ADVERSE EVENTS:
Description: Hyperkalemia in primary outcome is when patient experiences any AE after randomization with preferred term Hyperkalaemia or Blood potassium increased and AE table has incidences of AEs on or after randomization by preferred terms which exceeds a threshold of 2%. therefore 3 less cases than Primary OM.
Arm/Group | LCZ696 Condensed | LCZ696 Conservative
Serious Adverse Events (participants affected / at risk) | 21/246 | 14/251
Other Adverse Events (participants affected / at risk) | 72/246 | 52/251
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 Condensed (N=246) | LCZ696 Conservative (N=251)
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1
Cardiac failure (Cardiac disorders) | 3 | 2
Cardiac failure acute (Cardiac disorders) | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 1
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Cardiogenic shock (Cardiac disorders) | 3 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0
Coronary artery stenosis (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0
Ventricular tachycardia (Cardiac disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Cardiac death (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Hepatic cyst (Hepatobiliary disorders) | 1 | 0
Gastrointestinal infection (Infections and infestations) | 0 | 1
Infected skin ulcer (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 0
Staphylococcal sepsis (Infections and infestations) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Procedural complication (Injury, poisoning and procedural complications) | 0 | 1
International normalised ratio increased (Investigations) | 1 | 0
Bladder neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 2 | 0
Renal failure chronic (Renal and urinary disorders) | 1 | 0
Postmenopausal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 Condensed (N=246) | LCZ696 Conservative (N=251)
Cardiac failure (Cardiac disorders) | 6 | 1
Vertigo (Ear and labyrinth disorders) | 7 | 3
Nasopharyngitis (Infections and infestations) | 6 | 3
Hyperkalaemia (Metabolism and nutrition disorders) | 16 | 11
Hypokalaemia (Metabolism and nutrition disorders) | 6 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 2
Dizziness (Nervous system disorders) | 8 | 6
Renal failure (Renal and urinary disorders) | 2 | 7
Renal impairment (Renal and urinary disorders) | 10 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 6
Hypotension (Vascular disorders) | 24 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety.